CLINICAL TRIAL: NCT03960242
Title: Longitudinal Exploratory Prospective Evaluation of Clinical Evolution in Patients With Motor Predominant Parkinson Disease.
Brief Title: Evaluation of Clinical Progression in Patients With Motor Predominant Parkinson Disease.
Acronym: PARK001
Status: Terminated | Type: Observational
Why Stopped: Programs strategy refining due to Covid crisis
Sponsor: BrainEver (Industry)
Responsible Party: Sponsor
Other Study IDs: BREN01_CLIN_001
Record Dates: First submitted 2019-05-10; First posted 2019-05-23 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is the longitudinal prospective clinical evaluation in patients with motor predominant PD; it will assess the individual disease progression (change) of the clinical and imaging parameters measured at 6-month interval over a minimum of 12 months.

DETAILED DESCRIPTION:
The absence of clear PD subtypes defining a common path and rate of disease progression, combined with the absence of validated biomarkers indicative of disease progression and a strong placebo effect, constitute a challenge for clinical trials assessing new potential disease-modifying therapies in PD.

The present cohort would constitute a well-defined population of patients, with individual progression assessment, suitable to evaluate new disease-modifying therapies in a subsequent Phase1/2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's Disease (According to British Brain Bank Criteria); genetic forms of PD are not excluded
2. Male or female adult, aged 70 or less
3. Modified Hoehn and Yahr stage 2 to 3 in OFF state
4. Disease duration, i.e. time from first motor symptoms between 2 to 8 (included) years ; first motor symptoms to be taken into consideration being the cardinal motor symptoms of PD (bradykinesia, tremor and rigidity)
5. Univoqual response to L-DOPA (of at least 50% in MDS-UPDRS Part III motor score)
6. Presence of fluctuations and/or dyskinesia
7. MDS-UPDRS total motor score ≥15 in OFF state
8. L-Dopa treatment stable for at least 4 weeks
9. Covered by healthcare insurance
10. Written informed consent form signed

Exclusion Criteria:

1. Scan Without Evidence of Dopamine Deficit (SWEDD) (DaTSCAN)
2. Atypical parkinsonism syndrome
3. Dementia as detected by a score < 21/30 at the Montreal Cognitive Assessment Screening (MoCA)
4. Psychiatric disorders including major depression with suicidal thoughts as evaluated by a psychiatrist or a neurologist at the selection period
5. Any medical or psychological problems which may interfere with a smooth conduction of the study protocol (e.g. cancer with a limited life expectancy)
6. History of significant brain or vascular disease (tumor, epilepsy, stroke …)
7. Any contraindication for undergoing MRI of the head
8. Prior brain surgical procedures with or without implementation of an intra-cerebral device
9. Drug or alcohol addiction
10. Pregnancy or breastfeeding
11. Patient with reproductive potential who do not agree to use an accepted effective method of contraception - investigator's judgment- during the study period
12. Illiteracy or insufficient language skills (French) to complete the questionnaires
13. Patient deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection (e.g. guardianship or curatorship).
14. Simultaneous participation in another clinical trial with the administration of investigational drug(s)

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with motor predominant PD aged 70 or less, with a disease onset between 2-8 years.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS Part III) "off" medications | baseline, 6, 12, 18, 24 and 30 months after baseline ]
  An examiner will measure MDS-UPDRS part 3 motor scores "off" medications. MDS-UPDRS Part III is a motor examination consisting of 18 summed items where the investigator rates each motor symptom based on a scale of 0 - 4, higher values indicating worse function.

SECONDARY OUTCOMES:
Change from Baseline of brain MRI | 12 and 24 months
  neuromelanin sequence

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Pitié-Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: No